CLINICAL TRIAL: NCT07214285
Title: Evaluation of Long-term Safety in Parkinsonian Patients With Intracerebroventricular Administration of A-dopamine (Anaerobic Dopamine) DIVE-FOLLOW UP
Brief Title: Evaluation of Long-term Safety in Parkinsonian Patients With Intracerebroventricular Administration of A-dopamine (Anaerobic Dopamine)
Acronym: DIVE-FOLLOW UP
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: InBrain Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025_0243
Record Dates: First submitted 2025-09-25; First posted 2025-10-09 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- A-DOPAMINE (Experimental)
  Interventions: Drug: A-DOPAMINE; Device: A-DOPAMINE

INTERVENTIONS:
Drug: A-DOPAMINE — Intracerebral infusion of anaerobic dopamine.
Device: A-DOPAMINE — Intracerebral infusion of anaerobic dopamine with pump device.

SUMMARY:
Patients included in DIVE I have been receiving this treatment for several years as part of their participation in the study, which is scheduled to end on September 30, 2025. In this context, Lille University Hospital is offering patients still enrolled in DIVE I who wish to do so the opportunity to participate in a new clinical study, "Dive Follow Up," which is a longer-term follow-up study with, if necessary, a dose reduction until the experimental treatment is discontinued and an alternative treatment is put in place. It appears necessary to anticipate the discontinuation of treatment in order to limit as much as possible situations of abrupt discontinuation potentially associated with more severe clinical consequences. Thus, in order to limit the impact of discontinuing this treatment, the sponsor proposes a gradual and individualized reduction in the dose of A-dopamine and, whenever possible, an alternative treatment, in particular the new Scyova treatment.

The objective of this study will therefore be to monitor the safety of both long-term A-dopamine treatment and the consequences of discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the DIVE I study still being treated with A-dopamine.
* Social security beneficiary.
* Able to give free and informed consent to participate in the research.
* Patient willing to comply with all study procedures and duration.
* Patient not planning to change their lifestyle (nutritionally, physically, and socially) during their participation in the study.

Exclusion Criteria:

* Patients not included in DIVE I and not treated with A-dopamine.
* Presence of another serious condition that is life-threatening in the short or medium term, malnourished or cachectic patients.
* Taking treatments containing guanethidine or its relatives, or non-selective and selective monoamine oxidase A inhibitors (iproniazid, moclobemide, toloxatone)
* Patients already participating in another therapeutic trial involving the use of an experimental drug other than DIVE I or in an exclusion period
* Isolated patients, defined as those without a caregiver present for at least 3 hours/day at the patient's home

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events | Through study completion, an average of 1 year
  Recording of adverse events at any time. Frequency of adverse events reported by the patient and/or observed by the physician and/or home nurse during clinical examination, ECG, blood pressure, pulse, and standard laboratory tests.

CONTACTS AND LOCATIONS:
Locations (1):
- UHLillle, Lille, Haut de France, France